CLINICAL TRIAL: NCT06157398
Title: Diet Intervention Pilot: Refining a Meal and Food Delivery Approach
Acronym: FIRE-Diet-P
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Emily Brigham, Assistant Professor, University of British Columbia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: H22-02546
Record Dates: First submitted 2023-08-11; First posted 2023-12-05 (Actual); Last update posted 2024-11-27 (Actual); Status verified 2024-01

CONDITIONS: Healthy Individuals
Keywords: Diet Intervention; EPA; DHA; Omega-3 fatty acids
MeSH Terms: interventions — Fruit

STUDY DESIGN:
Intervention Model Description: 1. To inform feasibility and acceptability of the intervention for deployment in a future randomized control trial.
  2. Optimization of the design and implementation of a dietary intervention aimed at increasing intake of fruits, vegetables, and Omega-3 fatty acids in fish.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Diet Intervention (Other): Participants will be provided with a diet that has an increased intake of fish high in Omega-3 fatty acids as well as fruits and vegetables in comparison to their baseline intakes as assessed by the study dietician.
  Interventions: Other: Increased EPA, DHA, fruit, and vegetable intake

INTERVENTIONS:
Other: Increased EPA, DHA, fruit, and vegetable intake — Participants will receive food deliveries for approximately 4-weeks via online ordering, meal delivery, and dietician counseling.

SUMMARY:
A diet with a higher intake of fish and fruits, and vegetables, has shown promise in reducing inflammation and oxidative stress in the body. Intake of a diet with these components has been linked to fewer respiratory symptoms and lower rates of lung disease in multiple studies. In addition, emerging research suggests that a diet with these components may have the power to protect the body against some of the effects of exposure to air pollution.

In this study, participants will receive food, meals, and counseling designed to increase their dietary intake of fish, fruits, and vegetables. The research team will test the change in diet and learn ways to optimize the participants' experience.

DETAILED DESCRIPTION:
This study is anticipated to enroll up to 30 participants, who will be asked to complete a total of 3 visits to Vancouver General Hospital. The study will take at least 5 weeks to complete, and participants will be asked to dedicate about 11.5 hours of their time for the entire study, including 4 phone calls. The principal investigator may request to access their health records for medication or past medical history to ensure their safe participation in the study.

Participants will receive at least weekly home delivery of foods and meals to meet the nutritional goals of the dietary intervention, which include:

1. An average daily intake of 8-10 servings of fruits and vegetables high in antioxidants.

   To meet this goal, a study dietician will call participants weekly to assist in ordering fruits and vegetables of their choice that meet the needs of the study and assist them in some aspects of meal planning related to these orders. These fruits and vegetables will arrive by commercially-available grocery delivery.
2. An average daily intake of over 850 mg of omega-3 fatty acids (specifically eicosapentaenoic acid and docosahexaenoic acid, also known as EPA and DHA) from fish.

To meet these goals, the study dietician will also assist participants in ordering weekly, prepared, microwaveable meals from a meal delivery service. Participants will receive four fish meals per week, which will meet the requirements of this average daily intake; participants are not required to (nor is it necessary to) eat fish every day.

ELIGIBILITY:
Inclusion Criteria:

* Healthy: defined as no significant respiratory, cardiac, or metabolic disorders (e.g. obesity, diabetes)
* No dietary supplement use (vitamins, fish oil, etc.), or willing to stop the use of supplements for one month prior to study initiation and during the study period (if the supplement is prescribed or physician-recommended, the participant will be excluded from participation)
* No use of medications known to interact with diet composition (e.g. Coumadin)
* At the time of enrolment, consuming less than 250 mg EPA+DHA daily (<2 servings fish/week) and <5 servings of fruit/vegetables per day, assessed by dietary screeners
* Not actively participating in other studies that would provide conflict with this or the alternate study protocol

Exclusion Criteria:

* Pregnant or planning to become pregnant during the study period
* Actively attempting to lose weight
* Food allergies/intolerance or food aversion preventing adherence to the intervention diet, or unwillingness/medically unable to adjust diet in line with the intervention
* Plans to move outside of British Columbia during the study period
* Lack of access to adequate food storage or food preparation appliances

These inclusion and exclusion criteria align with the anticipated inclusion criteria for an upcoming diet and air pollution exposure study for which this pilot is informing the dietary intervention.

Ages: 19 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2024-01-29 (Actual); Primary Completion 2024-09-05 (Actual); Study Completion 2024-09-05 (Actual)

PRIMARY OUTCOMES:
Feasibility: Recruitment success | Through study completion (approximately 5 weeks/participant)
  Measures of recruitment success informing feasibility will include:
  Ratio of # in-person screens/# telephone pre-screening Ratio of # participants enrolled/# telephone pre-screening Ratio of # participants enrolled/# in-person screens
Feasibility: Protocol completion | Through study completion (approximately 5 weeks/participant)
  Measures of protocol completion informing feasibility will include:
  * participants completing visit 1
  * participants completing visit 2
  * participants completing visit 3

SECONDARY OUTCOMES:
Feasibility: Protocol adherence (dietary change) | From initiation of diet intervention to study completion (approximately 4 weeks/participant)
  Protocol adherence informing measurable change will be evaluated as follows:
  % completion of 24-hour recalls (6 planned per participant) Change in within-individual reported servings of fruit and vegetables across 4-week intervention (Wilcoxon matched pairs signed rank test) Change in within-individual reported servings of fish across 4-week intervention (Wilcoxon matched pairs signed rank test) Change in within-individual reported grams of omega-3 intake across initial 2 weeks and full 4-weeks of intervention (paired sample t-test) Change in blood biomarker (omega-3, carotenoid, LDL, HDL, total cholesterol) levels across initial 2 weeks and full 4-weeks of intervention (paired sample t-test)

OTHER OUTCOMES:
Acceptability of the Protocol | Through study completion (approximately 5 weeks/participant)
  Feedback provided at in-person visits 2 and 3 will be reviewed and described via qualitative interview. No formal statistical analysis is planned, and these results will be published.

CONTACTS AND LOCATIONS:
Overall Officials: Emily Brigham, MD, Principal Investigator — University of British Columbia
Locations (1):
- University of British Columbia, Vancouver, British Columbia, Canada